CLINICAL TRIAL: NCT05446753
Title: Singapore Healthy Alternative Protein Evaluation Study
Acronym: SHAPES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Prince September Pte. Ltd. (Unknown)
Responsible Party: Principal Investigator, JeyaKumar Henry, Deputy Executive Director, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022/00278
Record Dates: First submitted 2022-06-23; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases; Protein Metabolism Disorder
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases | interventions — Meat Substitutes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal-based meats (ABMD group) (Experimental): Participants will be instructed to substitute protein-rich foods consumed habitually with animal-based meats (ABMD group).
  Interventions: Dietary Supplement: Animal-based meats
- Plant-based meat alternatives (PBMD group) (Experimental): Participants will be instructed to substitute protein-rich foods consumed habitually with Plant-based meat alternatives (PBMD group).
  Interventions: Dietary Supplement: Plant-based meat alternatives

INTERVENTIONS:
Dietary Supplement: Animal-based meats — Animal-based meats from beef, pork and chicken
  Arms: Animal-based meats (ABMD group)
Dietary Supplement: Plant-based meat alternatives — Plant-based meat alternatives of beef, pork and chicken
  Arms: Plant-based meat alternatives (PBMD group)

SUMMARY:
The overall aim of this randomized controlled trial is to investigate the effects of consuming a Plant-Based Meat alternative Diet (PBMD) compared to an Animal-Based Meat Diet (ABMD) on cardiometabolic health and protein homeostasis in Chinese men and women in Singapore. This will be achieved through the following specific objectives: (1) To evaluate the effects of dietary protein source on metabolic health and glycemic control(2) To evaluate the effects of dietary protein source on risk factors of cardiovascular diseases (3) To evaluate the effects of dietary protein source on protein homeostasis and metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese males and females
2. Age > 30 to </= 70 years
3. Habitually consuming between 2 and 4 servings of protein-rich foods daily (~20 g protein per serving)
4. Raised blood glucose (fasting glucose >/= 5.4 and </= 7.0 mmol/L) and/or (HbA1c >/= 5.7 and </= 6.4 %)
5. Fully vaccinated against COVID-19 (referred to as having completed a minimum of 2 doses Pfizer-BioNTech / Comirnaty / Moderna or 3 doses Sinovac-CoronaVac)
6. Ability to give an informed consent
7. Willing to adhere to study intervention procedures

Exclusion Criteria:

1. Obese: BMI (>/= 27.5 kg/m2) and/or waist circumference (>/= 102 cm for male; >/= 88 cm for female)
2. Significant weight change (± 5 % body weight) during the past 3 months
3. Past bariatric surgery
4. Women who are pregnant, lactating or planning pregnancy
5. History or known present diagnosis of cardiovascular (i.e.hypertension (systolic/diastolic blood pressure: >/= 140/90 mmHg), endocrine (i.e. type 1 and type 2 diabetes mellitus), gastrointestinal, hematological (G6PD and coagulation disorders), hepatic (hepatitis B and C), malignant, renal, respiratory, thyroid or other relevant disorders which may affect the outcomes of interested in consultation with the researchers involved
6. Prescribed and regularly taking western or traditional medicine which may affect the outcomes of interest in consultation with the researchers involved
7. History or present diagnosis of HIV and/or tuberculosis.
8. Drug abuse within the last 5 years
9. Taking dietary supplements which may affect study outcomes one month prior to their first visit (e.g. protein supplements, omega-3/6 supplements or other nutritional supplements such as Ensure, Anlene etc.)
10. Following any special diets which may interfere with intervention procedures (for medical, aesthetic or religious reasons)
11. Allergy to nuts, seeds, legumes (soy, pea), cereal (wheat gluten), beef, pork, chicken or any other ingredients present in foods provided for intervention
12. Excessive alcoholic beverage consumption > 2 servings per day (1 serving is defined as 360 mL beer, 150 mL wine or 45 mL distilled spirits)
13. Smoking (cigarette, e-cigarette, cigar, pipe) or vaping
14. Exercising vigorously over the past 3 months
15. Staff of Prince September Pte. Ltd. (Pinduoduo Inc.) and/or Singapore Institute of Food and Biotechnology Innovation (SIFBI)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change in metabolic health risk indicators | Pre- and Post-intervention (Week 8)
  Glucose
Change in cardiovascular health risk indicators | Pre- and Post-intervention (Week 8)
  Insulin
Change in metabolic health risk indicators | Pre- and Post-intervention (Week 8)
  Fructosamine
Change in metabolic health risk indicators | Day -2 (from Week 0) to Day 12. 14 days in total
  14-day continuous blood glucose monitoring (subgroup; n = 48)
Change in cardiovascular health risk indicators | Pre- and Post-intervention (Week 8)
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglycerides
Change in cardiovascular health risk indicators | Pre- and Post-intervention (Week 8)
  Clinic blood pressure and ambulatory blood pressure (subgroup; n = 48)

SECONDARY OUTCOMES:
Change in protein metabolism-related biomarkers in plasma/serum | Pre- and Post-intervention (Week 8)
  Protein and amino acid profile
Change in protein metabolism-related biomarkers in plasma/serum | Pre- and Post-intervention (Week 8)
  Urea nitrogen
Change in protein metabolism-related biomarkers in plasma/serum | Pre- and Post-intervention (Week 8)
  Creatinine
Change in protein metabolism-related biomarkers in plasma/serum | Pre- and Post-intervention (Week 8)
  Albumin
Change in inflammation-related risk indicators | Pre- and Post-intervention (Week 8)
  High sensitivity CRP
Change in anthropometric measurements | Pre- and Post-intervention (Week 8)
  Weight
Change in anthropometric measurements | Pre- and Post-intervention (Week 8)
  Waist and hip circumference
Change in body composition | Pre- and Post-intervention (Week 8)
  Dual Energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toh DWK, Fu AS, Mehta KA, Lam NYL, Haldar S, Henry CJ. Plant-Based Meat Analogs and Their Effects on Cardiometabolic Health: An 8-Week Randomized Controlled Trial Comparing Plant-Based Meat Analogs With Their Corresponding Animal-Based Foods. Am J Clin Nutr. 2024 Jun;119(6):1405-1416. doi: 10.1016/j.ajcnut.2024.04.006. Epub 2024 Apr 8. PMID 38599522